CLINICAL TRIAL: NCT05977036
Title: BettER: Biomarker Driven Early Therapeutic Selection in Patients With HR+ HER2- Metastatic or Unresectable Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Biovica (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202307176
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer; Unresectable Breast Cancer
Keywords: ER+ HER2- metastatic breast cancer; biomarkers; thymidine kinase
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- TKa suppressed at Cycle 1 Day 15 (Experimental): * Study visits will occur at Baseline, Week 2 (C1D15), C2D1, C4D1, and clinical progression. Blood serum samples will be collected and analyzed using DiviTum® TKa at each of these dictated time points.
  * Patients with suppressed TKa levels at C1D15 will continue on CDK4/6i + endocrine therapy until clinical progression. There will be an option to elongate the time between restaging scans from Q3M to Q6M if TKa remains suppressed in this group. Physicians may repeat TKa in 2 weeks if TKa rise is noted and if TKa again becomes suppressed, may delay imaging. These patients will undergo TKa level monitoring at C2D1, C4D1, every 3 months thereafter, and at the time of clinical progression. The feasibility endpoint relates specifically to the Week 24 imaging time point.
  Interventions: Device: DiviTum® TKa assay; Drug: CDK4/6 + Endocrine therapy
- TKa unsuppressed at Cycle 1 Day 15 (Experimental): * Study visits will occur at Baseline, Week 2 (C1D15), C2D1, C4D1, and clinical progression. Blood serum samples will be collected and analyzed using DiviTum® TKa at each of these dictated time points.
  * Patients with lack of TKa suppression at C1D15 (defined as >145 DuA) will be recommended to switch to an alternative therapy after compliance with the medication is ensured (by pill count) and potential drug-drug interactions are reviewed. These patients will have TKa samples drawn at initiation of second-line therapy and on the first day of subsequent cycles until progression.
  Interventions: Device: DiviTum® TKa assay; Drug: CDK4/6 + Endocrine therapy
- Physicians (No Intervention): -Physicians will be asked to complete surveys as follows:
  * Physician Survey 1 for patients in the TKa C1D15 Suppressed group who have the option to delay the Week 24 scan at Week 24
  * Physician Survey 2 for patients in the TKa C1D15 Unsuppressed group at C1D15 (after TKa results have returned but before switching therapy)

INTERVENTIONS:
Device: DiviTum® TKa assay — Will be utilized for determination of serum enzymatic activity of TK1 according to the manufacturer's instructions
  Arms: TKa suppressed at Cycle 1 Day 15; TKa unsuppressed at Cycle 1 Day 15
Drug: CDK4/6 + Endocrine therapy — FDA-approved endocrine therapy plus CDK4/6 inhibitor. Ribociclib is the preferred CDK4/6 inhibitor. In the event this drug cannot be obtained due to insurance authorization or if there are specific side effect profile concerns from the treating physician, an alternative CDK4/6 inhibitor is allowed.
  Arms: TKa suppressed at Cycle 1 Day 15; TKa unsuppressed at Cycle 1 Day 15

SUMMARY:
This is a prospective study to assess the impact of biomarker driven, early therapeutic switching and delayed imaging with the incorporation of DiviTum® serum TK1 activity ("DiviTum® TKa") in patients with HR positive, HER-2 negative metastatic or unresectable breast cancer. Patients will receive first-line treatment with a CDK4/6 inhibitor (CDK4/6i) and endocrine therapy. All patients will have blood drawn for thymidine kinase activity (TKa) testing at baseline and at C1D15. Patients who are found to have a lack of TKa suppression at C1D15 will be recommended to switch to an alternative therapy. Patients with suppressed C1D15 TKa levels will continue on CDK4/6i and endocrine therapy until clinical progression. Patients with TKa which remains suppressed will be recommended to delay restaging scans from 24 weeks to 36 weeks.

The investigators hypothesize that a patient's TKa level at C1D15 is prognostic for progression-free survival (PFS) on a CDK4/6 inhibitor and early therapeutic switching in patients with a lack of C1D15 TKa suppression will be associated with prolonged PFS.

ELIGIBILITY:
Inclusion Criteria - Patients

* Diagnosis of metastatic or advanced unresectable invasive breast cancer that is hormone receptor-positive (HR+) and HER2-negative.
* Planned to initiate standard of care first-line therapy with FDA-approved endocrine therapy plus CDK4/6 inhibitor for the stated diagnosis at the time of study enrollment. Ribociclib is the preferred CDK4/6 inhibitor. In the event this drug cannot be obtained due to insurance authorization or if there are specific side effect profile concerns from the treating physician, an alternative CDK4/6 inhibitor is allowed.
* Any prior therapy for early stage breast cancer is allowed, including endocrine therapy and chemotherapy.
* Prior receipt of adjuvant CDK 4/6 inhibitor therapy is permitted provided therapy completion occurred > 12 months prior to study enrollment.
* Presence of RECIST-evaluable disease. Patients with bone-only disease are eligible.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Post-menopausal status, defined as one of the following:

  * Age ≥ 60 years
  * Age < 60 with intact uterus and amenorrhea for 12 consecutive months or more
  * Status post bilateral oophorectomy, total hysterectomy
  * Pre- or peri-menopausal with suppressed ovarian function by use of GnRH agonist/antagonist or surgical bilateral oophorectomy
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria - Patients

* Receipt of any prior cytotoxic chemotherapy line for metastatic disease. There will be no limit to chemotherapy use in the neoadjuvant or adjuvant setting.
* Patients with a prior or concurrent malignancy are excluded unless that malignancy's natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Concurrent participation in any investigational therapeutic trial for treatment of metastatic breast cancer.

Eligibility Criteria - Physicians

* Medical Oncologist at Siteman Cancer Center.
* Treating patients with metastatic or advanced unresectable breast cancer.
* Willing to complete Physician Surveys during participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2034-09-30 (Estimated); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in patients who remain on CKD4/6i (patients with suppressed TKa levels at cycle 1 day 15) | Through completion of follow-up (estimated to be 7 years)
  . PFS in patients with suppressed TKa levels is defined as from the start date of receiving CDK4/6i to the end date of CDK4/6i or last date on CDK4/6i if the treatment on CDK4/6i is still ongoing or date of death if death occurs on treatment.
Clinical benefit rate (CBR) in patients who remain on CDK4/6i | Through completion of follow-up (estimated to be 7 years)
  CBR is defined as total number (or percentage) of patients who achieved a complete response, partial response, or had stable disease for 6 months or more.
Progression-free survival (PFS) in patients who switch to an alternate therapy (patients with unsuppressed TKa levels at cycle 1 day 15) | Through completion of follow-up (estimated to be 7 years)
  PFS in patients with unsuppressed TKa levels is defined as from the start date of receiving CDK4/6i to the end date of next-line therapy or last date on next-line if the treatment on next-line therapy is still ongoing or date of death if death occurs on treatment.

SECONDARY OUTCOMES:
Feasibility (compliance rate) in patients with suppressed TKa level at cycle 1 day 15 | At 36 weeks
  -Feasibility defined as compliance rate:
  **Patients with suppressed TKa at C1D15, C2D1, C4D1 and 24 weeks: compliance is defined as this subset of physicians and patients who delay restaging scans from 24 weeks to 36 weeks.
Feasibility (compliance rate) in patients with unsuppressed TKa level at cycle 1 day 15 | At Cycle 1 Day 15
  -Feasibility defined as compliance rate:
  **Patients with unsuppressed TKa at C1D15: compliance is defined as subset of physicians and patients following protocol recommendation to switch to next line of treatment.
Baseline TKa level to predict overall survival (OS) on first-line CDK4/6i | Through completion of follow-up (estimated to be 7 years)
  OS is defined as from the start date of receiving CDK4/6i to the date of death or date of last follow up.
Baseline TKa level to predict overall survival (OS) on later lines of therapy | Through completion of follow-up (estimated to be 7 years)
  OS is defined as from the start date of receiving CDK4/6i to the date of death or date of last follow up.
Cycle 1 day 15 TKa level to predict overall survival (OS) on first-line CDK4/6i | Through completion of follow-up (estimated to be 7 years)
  OS is defined as from the start date of receiving CDK4/6i to the date of death or date of last follow up.
Cycle 1 day 15 TKa level to predict overall survival (OS) on later lines of therapy | Through completion of follow-up (estimated to be 7 years)
  OS is defined as from the start date of receiving CDK4/6i to the date of death or date of last follow up.
Cycle 2 day 1 TKa level to predict overall survival (OS) on first-line CDK4/6i | Through completion of follow-up (estimated to be 7 years)
  OS is defined as from the start date of receiving CDK4/6i to the date of death or date of last follow up.
Cycle 2 day 1 TKa level to predict overall survival (OS) on later lines of therapy | Through completion of follow-up (estimated to be 7 years)
  OS is defined as from the start date of receiving CDK4/6i to the date of death or date of last follow up.
Number of patients with TKa suppressed at cycle 1 day 15 who have stable disease on subsequent disease assessments | Through 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Clifton, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu